CLINICAL TRIAL: NCT03939754
Title: Dedalo Study Protocol: the Evaluation of a Community-level Multicomponent Lifestyle Intervention Effectiveness
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Responsible Party: Sponsor
Other Study IDs: AslVC.Med.18.02
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Lifestyle Risk Reduction
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult attendance to Dedalo activities: Adult attended one Dedalo's activity
  Interventions: Behavioral: Dedalo project
- Adult living in Vercelli: Adult aged 40-75

INTERVENTIONS:
Behavioral: Dedalo project — Physical activity, healthy food, socialization and mental activity promotion
  Groups: Adult attendance to Dedalo activities

SUMMARY:
The reduction of non-transmissible diseases (NCDs) is a community health priority and many NCDs are lifestyle related. In order to promote healthy lifestyle in Vercelli, the Local Health Authority (ASL) and the municipality of Vercelli and the University of Novara have realized the Dedalo project: a multicomponent community intervention. In Italy, few are the study evaluating the effectiveness of the multicomponent community intervention. Thus, aim of the study is to evaluate the effectiveness of Dedalo project in promoting lifestyle healthier change in the adult lifestyle general population in Vercelli.

DETAILED DESCRIPTION:
BACKGROUND. The reduction of the non-transmissible diseases (NCDs) is a priority for the health community and for the economical sustainability of the healthcare system. In fact, the NCDs are the main global cause of death. It is demonstrated that many NCDs are lifestyle related; notable, even small lifestyle changes bring a health outcome improvement. The Italian epidemiological survey PASSI (2013-2016) reveals that the 33% of the population aged 50-69 years old living in Vercelli is self-declared sedentary and the 45% is overweight/obese. The Dedalo project, started in March 2018, is finalized to promote evidence-based healthy behaviors in the Vercelli adult population. In Italy the studies of community multicomponent prevention interventions are few. In this regard, the aim of the study is to evaluate the Dedalo project efficacy in the promotion of lifestyle changes.

MATERIALS AND METHODS. The study is a prospective observational one. The socio-economical and behaviors information are detected through an ad hoc questionnaire. The questionnaire is telephone-administered to the population who attended Dedalo activities and to an adult general population sample (40-75 years old) living in Vercelli. The same questionnaire will be administered 12 months later the first interview.

EXPECTED RESULTS. In April 2018 the socio-economics and behaviors description of both the studied population will be available. The fist evaluation of behavioral change will be concluded in April 2019.

CONCLUSIONS. The study will allow to define the efficacy of the community prevention intervention Dedalo is behavioral changes promotion, its capability in involving all the target population promoting equality in health and to improve the community prevention interventions.

ELIGIBILITY:
Inclusion Criteria:

* adult population living in Vercelli municipality

Exclusion Criteria:

* inability to understand the Italian language
* inability to answer to the telephonic interview
* denial of the informed consent

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population living in Vercelli municipality aged 40-75 years old. The cohort consists in two sample: 214 person who attended at least one Dedalo activity, 214 person randomly selected from the ASL register of Vercelli.
Sampling Method: Probability Sample
Enrollment: 428 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the intervention effectiveness in promoting healthy lifestyle | 12 month (April 2019 - April 2020)
  Lifestyle habits detection and description through a telephone-based questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Faggiano, Study Chair — Eastern Piedmont University
Locations (1):
- Università degli Studi del Piemonte Orientale "Amedeo Avogadro", Novara, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hobbs N, Godfrey A, Lara J, Errington L, Meyer TD, Rochester L, White M, Mathers JC, Sniehotta FF. Are behavioral interventions effective in increasing physical activity at 12 to 36 months in adults aged 55 to 70 years? A systematic review and meta-analysis. BMC Med. 2013 Mar 19;11:75. doi: 10.1186/1741-7015-11-75. PMID 23506544
- [Background] Lawton BA, Rose SB, Elley CR, Dowell AC, Fenton A, Moyes SA. Exercise on prescription for women aged 40-74 recruited through primary care: two year randomised controlled trial. BMJ. 2008 Dec 11;337:a2509. doi: 10.1136/bmj.a2509. PMID 19074218
- See also: Italian surveillance of behavioral risk factors — http://www.epicentro.iss.it/passi/